CLINICAL TRIAL: NCT05368493
Title: Prenatal Air Pollution and Neurodevelopment: a Longitudinal Neuroimaging Study of Mechanisms and Early Risk for ADHD in Puerto Rican Children
Brief Title: Air Pollution and Development in the Boricua Youth Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of Puerto Rico (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Claudia Lugo-Candelas, Assistant Professor, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8232; R01ES032870-01 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pollution; Exposure; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants will be in the same arm.
  Interventions: Other: MRI task

INTERVENTIONS:
Other: MRI task — Task fMRI (Simon) [ Time Frame: Children will undergo MRI scans when they are 6-11 years of age. ] Children will also complete a task, which will allow exploratory analyses of the functionality of attention-related neural circuits. The Simon fMRI task is a non-verbal task equivalent to the Stroop that tests sustained attention and inhibitory control and discriminates children with and without ADHD. Exploratory fMRI time-series data for each participant will be modeled using a general linear model with 3 predictors: congruent correct, incongruent correct, and incorrect. Contrast images for each participant (e.g., incongruent-minus-congruent) will be generated and entered into a group-level random-effects model. Analyses are exploratory, and will focus on frontal lobe activity during each type of trial.

SUMMARY:
This study seeks to understand the relationship between prenatal maternal air pollution exposure and offspring risk for ADHD and examine two potential -modifiable- mechanisms: prenatal maternal inflammation and offspring sleep problems. We will employ a longitudinal neuroimaging study design and leverage a well-characterized intergenerational cohort of Puerto Ricans to address prior literature's limitations. This will be the first study to use infant neuroimaging to disassociate the effects of prenatal pollution exposure from those of postnatal pollution exposure, adversity and disadvantage, and offspring genetic risk for ADHD.

DETAILED DESCRIPTION:
The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June, 2023.

The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Having been enrolled in the BYS-ECHO birth cohort (parent study).
* Speaks English or Spanish.
* Having a parent that is eligible to participate, based on criterial detailed below, and agrees to participation.
* One parent must speak English or Spanish.

Exclusion Criteria:

* Having serious neurological disorder, excluding ASD (e.g., seizure disorder).
* MRI contraindications (irremovable metal in body like braces, pacemakers).
* Claustrophobia.
* Having a parent that is not competent to consent (e.g., severe intellectual disability would have triggered exclusion) or under 18 years of age.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Frontal lobe and corpus callosum volumes | Children will be scanned either at 6-36 months or 6-11 years of age, depending on when the participants are enrolled.
  Frontal lobe and corpus callosum volumes in will be measure in offspring. Bilateral middle frontal cortex and corpus callosum volumes will be used in hypothesis testing.

OTHER OUTCOMES:
Exploratory- Task fMRI (Simon) | Children will undergo MRI scans when they are 6-11 years of age.
  Children will also complete a task, which will allow exploratory analyses of the functionality of attention-related neural circuits. The Simon fMRI task is a non-verbal task equivalent to the Stroop that tests sustained attention and inhibitory control and discriminates children with and without ADHD. Exploratory fMRI time-series data for each participant will be modeled using a general linear model with 3 predictors: congruent correct, incongruent correct, and incorrect. Contrast images for each participant (e.g., incongruent-minus-congruent) will be generated and entered into a group-level random-effects model. Analyses are exploratory, and will focus on frontal lobe activity during each type of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia I Lugo-Candelas, PhD, Principal Investigator — Columbia University Irving Medical Center/New York State Psychiatric institute; Glorisa Canino, PhD, Principal Investigator — University of Puerto Rico; Cristiane S Duarte, PhD, Principal Investigator — Columbia University Irving Medical Center/New York State Psychiatric institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant level data will be shared as required by NIH's 2003 Data Sharing Policy. The data sharing plan and elements are still being determined.